CLINICAL TRIAL: NCT05501574
Title: An Open Label Trial Evaluating the Safety, Tolerability, Efficacy and Pharmacokinetic Profile of Tacrolimus Inhalation Powder in Adult Lung Transplant Recipients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to funding constraints
Sponsor: TFF Pharmaceuticals, Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TFF-T2-001
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Lung Transplant Rejection
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Tacrolimus Inhalation Powder (Experimental): Single arm open label
  Interventions: Drug: Tacrolimus Inhalation Powder; Device: Plastiape RS00 Dry Powder inhaler device

INTERVENTIONS:
Drug: Tacrolimus Inhalation Powder — Tacrolimus powder for inhalation to prevent acute allograft rejection
  Other Names: Tacrolimus
Device: Plastiape RS00 Dry Powder inhaler device — dry powder inhaler device

SUMMARY:
Part A: This is an open label, single-arm study that will evaluate the safety, tolerability, efficacy and PK of Tacrolimus Inhalation Powder over 12 weeks in lung transplant patients who require reduced blood levels of tacrolimus due to kidney toxicity. Tacrolimus Inhalation Powder is being developed as an alternative to oral tacrolimus for prevention of rejection in adult lung transplant recipients.

Part B of this study is an optional safety extension following successful completion of Part A. Patients would have the option to continue Tacrolimus Inhalation Powder for up to 1 year, with a possibility to extend to 2 years pending analysis of Part A data. Participants would return to clinic every 12 weeks for safety assessments, dose adjustments, and to receive more Tacrolimus Inhalation Powder. After 2 years, if the drug is still under development, the subject will be invited to continue receiving Tacrolimus Inhalation Powder under a special access program.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent to participate and is willing and able to participate in the study and abide by study restrictions in the judgement of the Investigator.
2. Males or females aged 18 or over at time of screening.
3. Continuous non-smoker who has not used nicotine-containing products (including e-vaping) for at least 12 weeks prior to the first dosing and throughout the study, based on patient's self-reporting and urine cotinine levels at screening and Day 1.
4. Have undergone bilateral allograft lung transplantation at least six months prior to enrolment and meet all of the following:

   1. Receiving oral immediate-release or oral extended-release (not intravenous [IV] or sublingual) tacrolimus immunosuppression at a stable dose for 3 weeks prior to first dosing according to institutional standards as part of an immunosuppressive regimen along with mycophenolate mofetil or azathioprine and corticosteroids
   2. Demonstrating elevated markers of renal dysfunction: blood serum creatinine > 124 μmol/L (0.14 mg/dL) or estimated glomerular filtration rate (eGFR) < 45
   3. Stable to enable routine post-treatment bronchoscopy with BAL and EBB. Biopsy is not required in patients with significant increased risk of bleeding after Sponsor Medical Monitor approval.
   4. Screening FEV1 and forced vital capacity (FVC) values ≥ 40% predicted (to assure viable graft)
5. Females (women) of child-bearing potential (WOCBP) are defined as those who have experienced menarche and who have not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and who are not post-menopausal. WOCBP must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Day 1 and must agree to practice contraception as defined below if sexually active with males. In addition, no WOCBP may be planning a pregnancy during the study period.

   1. Female subjects who are WOCBP must agree to use highly effective contraceptive methods or abstinence for the duration of time on the study and continue to use acceptable contraceptive methods for 3 months after administration of the last dose of study treatment. Highly effective contraception is defined as use of the 2-barrier method (e.g., female diaphragm and male condom), 1 barrier method with spermicide, intrauterine device, or hormonal contraceptives (e.g., implant or oral). If the subject is using a hormonal form of contraception, use must have been stable for at least 4 weeks prior to screening.
   2. Abstinence will be acceptable only if it is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation) and withdrawal are not acceptable methods of contraception.
   3. Post-menopausal females are eligible if they meet the definition of menopause (at least 12 months of amenorrhea in the absence of other biological causes) and for females < 55 years of age, must also have a documented serum follicle stimulating hormone (FSH) level of > 40mIU/mL at Screening.
6. Male subjects with female partners of childbearing potential must be congenitally sterile or surgically sterile (vasectomy with confirmation of aspermia) or agree to use 2 effective methods of contraception including 1 barrier method (e.g., condom with spermicide and contraception by female partner) for the duration of time on the study and for 3 months after administration of the last dose of study treatment. Use of a condom is required by men during intercourse with a male or female partner to prevent potential delivery of the drug via seminal fluid during the study until the end of treatment visit.
7. If male, must agree not to donate sperm from the first dosing until 90 days after the last dosing.
8. Able to successfully perform spirometry, use the inhalation device, and comply with study restrictions and visit schedule.

Exclusion Criteria:

1. Active antibody-mediated rejection (AMR) or any other evidence of acute rejection
2. Active bacterial, viral or fungal infection not successfully resolved at least 4 weeks prior to study entry.
3. Presence of uncontrolled gastro-esophageal reflux disease (GERD)
4. History or presence of hypersensitivity or idiosyncratic reaction to tacrolimus or any calcineurin inhibitor.
5. Received a treatment with other investigational drug within 5 times the elimination half-life, if known (e.g., a marketed product) or within 30 days (if the elimination half-life is unknown), whichever is longer, prior to Study Day 1 dosing.
6. Positive for hepatitis B surface antigen (HBsAg) PCR, hepatitis C PCR, and human immunodeficiency virus (HIV) I and II antibodies, tuberculosis (TB), or COVID-19 at Screening.
7. Patients who have taken any of the following prohibited medications within 30 days of the first dose or who are expected to require these medications during the study:

   1. Cyclosporin
   2. Any form of sirolimus or everolimus
8. Allergy or sensitivity to lactose or milk products.
9. Clinically significant hepatic impairment defined as 5 times the upper limit of normal (ULN) for ALT and AST.
10. Patients receiving haemodialysis or peritoneal dialysis
11. Active post-transplant lymphoproliferative disorder (PTLD) related to Epstein-Barr Virus (EBV) infection.
12. Subjects with significant electrocardiogram (ECG) abnormalities at screening, including a QT interval corrected by the Fridericia correction formula that is ≥ 440 msec in men and ≥ 460 msec in women.
13. Demonstrates an inability to operate the inhalation device after training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Effect on renal function | Baseline through 12 weeks
  Mean change from baseline in renal function (glomerular filtration rate and creatinine) over time.
Incidence of treatment-emergent AEs, serious adverse events (SAEs), and withdrawals due to AEs. | baseline through 12 weeks
  safety and tolerability
Change in systolic and diastolic blood pressure (mm Hg) over time | baseline through 12 weeks
  safety and tolerability
Changes from baseline in potassium (mEq/L) over time | baseline through 12 weeks
  safety and tolerability
Changes from baseline in forced expiratory volume in one second (FEV-1) in liters | baseline through 12 weeks
  safety and tolerability
Changes from baseline in chest radiography | baseline through 12 weeks
  safety and tolerability
Number of participants with changes from baseline in physical examinations | baseline through 12 weeks
  safety and tolerability
Proportion of patients meeting treatment stopping rules. | baseline through 12 weeks
  safety and tolerability
Incidence of all-cause mortality and allograft-related mortality. | baseline through 12 weeks
  safety and tolerability
Incidence of all-cause hospitalization and allograft-related hospitalization | baseline through 12 weeks
  safety and tolerability
Efficacy of Tacrolimus Inhalation Powder in preventing acute rejection events | Baseline through 12 weeks
  Proportion of patients with no evidence of allograft rejection.
Efficacy of Tacrolimus Inhalation Powder in preventing acute rejection events | Baseline through 12 weeks
  Median time to first evidence of rejection.
Tacrolimus maximum concentration (Cmax) by visit | baseline through 12 weeks
  Pharmacokinetics
Tacrolimus time to maximum concentration (Tmax) by visit | baseline through 12 weeks
  Pharmacokinetics
Tacrolimus area under the curve from 0 to 6 hours (AUC0-6) by visit. | baseline through 12 weeks
  Pharmacokinetics
Tacrolimus area under the curve to last measurement (AUClast) by visit. | baseline through 12 weeks
  pharmacokinetics
Therapeutic drug monitoring tacrolimus blood levels by visit | baseline through 12 weeks
  Pharmacokinetics

SECONDARY OUTCOMES:
Blood and BAL biomarkers | Baseline through 12 weeks
  Ratio of BAL:Blood tacrolimus trough levels at Visit 1b and Visit 9b after oral and inhaled administration, respectively, and change in ratio.
DSA | Baseline through 12 weeks
  Donor-specific antibody levels (DSA) at baseline on oral tacrolimus and after treatment with Tacrolimus Inhalation Powder.
Acute allograft rejection from EBB samples | Baseline through week 12
  To determine if Tacrolimus Inhalation Powder reduces (if elevated) or maintains (if already low) signs of acute allograft rejection from endobronchial biopsy (EBB) samples compared with baseline oral tacrolimus therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zamaneh Mikhak, MD, Study Director — TFF Pharmaceuticals
Locations (2):
- Australia (2):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - The Alfred Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No